CLINICAL TRIAL: NCT00522912
Title: A Randomised Controlled Trial of Epilation Verses Immediate Surgery for the Management of Minor Trachomatous Trichiasis
Brief Title: A Trial of Epilation Verses Surgery for Minor Trichiasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5024
Record Dates: First submitted 2007-08-28; First posted 2007-08-30 (Estimated); Last update posted 2012-01-12 (Estimated); Status verified 2012-01

CONDITIONS: Trachomatous Trichiasis
Keywords: Trachoma; Trichiasis; Surgery; Epilation; Ethiopia
MeSH Terms: conditions — Trachoma; Trichiasis | interventions — Hair Removal

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Immediate posterior lamella tarsal rotation surgery for minor trichiasis
  Interventions: Procedure: Trichiasis surgery
- B (Active Comparator): Regular epilation by another person
  Interventions: Procedure: Epilation

INTERVENTIONS:
Procedure: Trichiasis surgery — Posterior lamella tarsal rotation
  Arms: A
Procedure: Epilation — Epilation of lashes by another well sighted person using quality epilating forceps
  Arms: B

SUMMARY:
Trachoma is the leading infectious cause of blindness worldwide. Recurrent infection by Chlamydia trachomatis causes a gradual scarring process of the inner surface of the eyelid (conjunctiva) leading to in-turning of the eyelids (entropion) and lashes touching the eye (trichiasis). The rate of progression and the severity of disease are variable. Some people develop severe disease with extensive entropion and trichiasis, whilst others have a mild problem with only a few lashes touching the eye, which does not progress.

In more advanced cases there is a broad consensus that the entropion / trichiasis should be corrected by surgery. In mild cases (minor trichiasis: 1-5 lashes touching the eye) the optimal treatment is uncertain. Some advocate early surgery to turn the eyelid out for any individual with one or more lashes touching any part of the eye. Others consider this to be too early for surgical intervention, as surgery can have a high recurrence rate and complications can arise. Instead, they recommend that minor trichiasis can be managed by epilation (pulling out lashes with forceps). In many endemic regions the uptake of surgery is low, with many patients preferring to epilate for mild disease.

The primary purpose of this study is to compare the outcome of immediate surgery to regular epilation for the management of minor trichiasis. The epilation would be done by a person with good eyesight using proper epilation forceps.

ELIGIBILITY:
Inclusion Criteria:

* Minor trichiasis: 1 - 5 lashes touching the eye

Exclusion Criteria:

* Previous eyelid surgery.
* Patients with evidence of corneal damage (will be offered surgery).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1300 (Actual)
Dates: Start 2008-03; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Trichiasis | One and two years

SECONDARY OUTCOMES:
Visual acuity | One and two years
Corneal opacity | One and two years

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J Burton, PhD FRCOphth, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (1):
- Bahir Dar Regional Health Bureau, Bahir Dar, Amhara, Ethiopia

REFERENCES:
- [Result] Rajak SN, Habtamu E, Weiss HA, Kello AB, Gebre T, Genet A, Bailey RL, Mabey DC, Khaw PT, Gilbert CE, Emerson PM, Burton MJ. Surgery versus epilation for the treatment of minor trichiasis in Ethiopia: a randomised controlled noninferiority trial. PLoS Med. 2011 Dec;8(12):e1001136. doi: 10.1371/journal.pmed.1001136. Epub 2011 Dec 13. PMID 22180731
- [Derived] Gower EW, Munoz B, Rajak S, Habtamu E, West SK, Merbs SL, Harding JC, Alemayehu W, Callahan EK, Emerson PM, Gebre T, Burton MJ. Pre-operative trichiatic eyelash pattern predicts post-operative trachomatous trichiasis. PLoS Negl Trop Dis. 2019 Oct 7;13(10):e0007637. doi: 10.1371/journal.pntd.0007637. eCollection 2019 Oct. PMID 31589610
- [Derived] Rajak SN, Habtamu E, Weiss HA, Bedri A, Zerihun M, Gebre T, Gilbert CE, Emerson PM, Burton MJ. Why do people not attend for treatment for trachomatous trichiasis in Ethiopia? A study of barriers to surgery. PLoS Negl Trop Dis. 2012;6(8):e1766. doi: 10.1371/journal.pntd.0001766. Epub 2012 Aug 28. PMID 22953007
- See also: Published Results — http://www.plosmedicine.org/article/info%3Adoi%2F10.1371%2Fjournal.pmed.1001136